CLINICAL TRIAL: NCT04569994
Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneous NNC0363-0845 in Healthy Subjects and in Subjects With Type 1 Diabetes
Brief Title: A Study to Look at the Safety of NNC0363-0845 in Healthy People and People With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1845-4598; U1111-1244-4315 (Other: World Health Organization (WHO)); 2019-004658-27 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Healthy Volunteers; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec

STUDY DESIGN:
Intervention Model Description: Part 1 will be a placebo-controlled trial in healthy subjects; Part 2 will be an active-controlled trial in subjects with T1D.
  Part 3 of this trial, will be an open-label, two-period cross-over, randomised, single dose trial in subjects with T1D.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Healthy volunteers will receive either NNC0363-0845 or placebo
  Interventions: Drug: NNC0363-0845; Drug: Placebo (NNC0363-0845)
- Part 2 (Experimental): Participants with T1D will receive either NNC0363-0845 or insulin degludec
  Interventions: Drug: NNC0363-0845; Drug: Insulin degludec
- Part 3 (Experimental): Participants with T1D will receive NNC0363-0845
  Interventions: Drug: NNC0363-0845

INTERVENTIONS:
Drug: NNC0363-0845 — A single dose administered s.c. (subcutaneously, under the skin)
Drug: Placebo (NNC0363-0845) — A single dose administered s.c.
  Arms: Part 1
Drug: Insulin degludec — A single dose administered s.c.
  Arms: Part 2

SUMMARY:
This study is investigating the safety and tolerability of the new investigational product NNC0363-0845, its concentrations in the blood and its effect on the blood sugar for the treatment of diabetes. The study consists of 3 parts. The first part of the study is conducted in healthy people, while the second part involves people with type 1 diabetes (T1D). Part 3 of this trial involves also people with T1D.

The study will test how NNC0363-0845 is tolerated by the body, how it is taken up in the blood, how long it stays there and how much the blood sugar is lowered. Healthy volunteers will either get NNC0363-0845 or placebo - which treatment is decided by chance. Participants with type 1 diabetes will either get NNC0363-0845 or insulin degludec (Tresiba®), also decided by chance. It is the first time that NNC0363-0845 is tested in humans. Participants will get one dose of NNC0363-0845 or placebo or insulin degludec injected into their left thigh. Participation in the study will last for up to 6 weeks. There will be one Informed Consent visit and 6 clinic visits with the study doctor. Healthy volunteers will have blood sampling to measure blood sugar and the concentration of the investigational product in the blood. Participants with type 1 diabetes will have a clamp experiment where the blood sugar is measured and controlled for up to 42 hours.

For Part 3, the total duration of the trial for each individual is expected to be approximately 3-9 weeks.

Participants cannot be in the study if the study doctor thinks that there are risks for their health. Women can only take part in the study if they are of non-child bearing potential.

ELIGIBILITY:
Inclusion Criteria:

Part 1 (healthy subjects):

* Male subject or female subject of non-child bearing potential. Non-child bearing potential being defined as surgically sterilised (i.e. documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or being postmenopausal (defined as no menses for 12 months without an alternative medical cause) prior to the day of screening.
* Aged 18-55 years (both inclusive) at the time of signing informed consent.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Part 2 and 3 (subjects with type 1 diabetes mellitus):

* Male subject or female subject of non-child bearing potential. Non-child bearing potential being defined as surgically sterilised (i.e. documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or being postmenopausal (defined as no menses for 12 months without an alternative medical cause) prior to the day of screening.
* Aged 18-55 years (both inclusive) at the time of signing informed consent.
* Diagnosed with type 1 diabetes mellitus 1 year or more prior to the day of screening.
* Glycated haemoglobin (HbA1c) equal to or below 8.5%.
* Fasting C-peptide below 0.30 nmol/L.
* Considered to be generally healthy (except for type 1 diabetes mellitus and sequelae of diabetes which may only be of mild severity) based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

Part 1 (healthy subjects) Part 2 and Part 3 (subjects with type 1 diabetes mellitus):

- Male of reproductive age who or whose partner(s) is not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice). Adequate contraceptive measures include that the male subject uses a condom during intercourse and that the partner practices adequate contraception (risk of pregnancy must be lower than 1%). In addition, subjects must not donate sperm for the duration of the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (AEs) | Part 1 and 2: From trial product administration at Visit 2, day 1 until completion of post treatment end-of-trial visit at Visit 6, day 10
  Number of events
Number of treatment-emergent adverse events (AEs) | Part 3: From trial product administration at Visit 2, day 1 until completion of post treatment end-of-trial visit at Visit 4 (up to 33 days after Visit 2, day 1)
  Number of events

SECONDARY OUTCOMES:
Number of treatment-emergent hypoglycaemic episodes | Part 1 and 2 From trial product administration at Visit 2, day 1 until completion of post treatment end-of-trial visit at Visit 6, day 10
  Number of episodes
Number of treatment-emergent hypoglycaemic episodes | Part 3: From trial product administration at Visit 2, day 1 until completion of post treatment end-of-trial visit at Visit 4 (up to 33 days after Visit 2, day 1)
  Number of episodes
Area under the serum NNC0363-0845 concentration-time curve from 0 to infinity after a single dose | Part 1 and 2 From 0 hours until last measurement time after trial product administration (Visit 2, day 1)
  pmol*h/L
Area under the serum NNC0363-0845 concentration-time curve from 0 to infinity after a single dose | Part 3: From 0 hours until last measurement time after trial product administration (Visit 2, day 1 and Visit 3, day 1)
  pmol*h/L
Maximum observed serum NNC0363-0845 concentration after a single dose | Part 1 and 2 From 0 hours until last measurement time after trial product administration (Visit 2, day 1)
  pmol/L
Maximum observed serum NNC0363-0845 concentration after a single dose | Part 3: From 0 hours until last measurement time after trial product administration (Visit 2, day 1 and Visit 3, day 1)
  pmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency and Medical Writing Office (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Mainz, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com